CLINICAL TRIAL: NCT00466414
Title: Alveolar Ridge Preservation With Polycaprolactone Scaffold for Implant Site Development
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-222-000-024-112
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2008-05

CONDITIONS: Alveolar Ridge Resorption After Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Polycaprolactone Scaffold

SUMMARY:
It has been shown through research that alveolar ridges (Part of jaw bone holding teeth) tend to lose width and height after extraction of teeth. Lost in height and width of the ridge can cause problems in the restoration of missing teeth with bridges and implants. Hence, this study is proposed to assess the use of polycaprolactone (PCL) scaffolds for alveolar ridge preservation following extraction of teeth in humans.

20 patients will be divided into 2 groups. In one group, patients will have a PCL scaffold placed into the socket after extraction. In other group, no scaffold will be placed. After a healing period of 6 months, changes in width and height from baseline is measured for both groups. A bone biopsy is also taken at this time from both groups. Hardness of bone, histologic (microscopic) features of cells, percentage of living bone, radiographic density of alveolar ridge and mechanical properties of the bone biopsy are then assessed.

This study will attempt to show that a resorbable (can be removed by body) material like a PCL scaffold can be used to maintain physical dimensions of the alveolar ridge after extraction and will not interfere with osseointegration (fusion with bone). It will avoid the necessity for additional corrective surgeries for patients when alveolar ridges presented with inadequate width and height for placement of aesthetically pleasing and functionally sound restorations. This would improve chances of success for the patient.

If the study successfully shows that the PCL scaffold can be accepted by the body with good bone growth, uses for the PCL scaffold can be extended to other areas of clinical medicine and dentistry.

The PCL scaffold to be used in this study is designed and developed by a local company (Osteopore International Pte Ltd). With the success of this product, Singapore's standing as a biomedical hub will be further enhanced.

ELIGIBILITY:
Inclusion Criteria:

1. Having 1 or more unsalvageable non-molar teeth indicated for extraction due to periodontal disease, endodontic failures, crown/root fractures, extensive caries or trauma
2. Have the indications for dental implant placement
3. Given alternative options and chose replacement by endosseous implants following extractions
4. If more than 1 tooth is to be replaced with implants, they should not be adjacent to each other
5. Position of unsalvageable tooth is close to final implant position
6. Good to fair oral hygiene (No probing depths <5mm and Gingivitis score of <20%)

Exclusion Criteria:

1. Immunocompromised state
2. Prior radiotherapy to extraction site
3. Chemotherapy in the past 12 months
4. Blood disorders
5. Uncontrolled diabetes
6. Uncontrolled hypertension
7. Long term steroid or anti-inflammatory therapy
8. Require antibiotic prophylaxis before dental treatment
9. Other uncontrolled systemic disease
10. Drug or alcohol abusers
11. Active infection in extraction site
12. Heavy smoker (> 10 sticks a day)
13. Pregnancy/Lactation
14. Known allergies to plastics or other polymer
15. Unwillingness to undergo basic dental treatment like caries-control and periodontal therapy
16. Failure to sign informed consent form

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03-12 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
To test the effectiveness of the PCL scaffold in maintaining the physical dimensions of the alveolar ridge after extraction.

SECONDARY OUTCOMES:
To assess the percentage of living bone that is formed during healing with presence of PCL scaffold.
To assess the possibility of using density of CT scan to determine the percentage of living bone in the site for implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Ang Chee Wan, BDS, Principal Investigator — National University of Singapore; Lim Thiam Chye, FRCS, Principal Investigator — National University Hospital, Singapore; Lim Lum Peng, MSc, Principal Investigator — National University of Singapore; Chung Kong Mun, MS, Principal Investigator
Locations (1):
- National University Hospital, Singapore, Singapore